CLINICAL TRIAL: NCT05768035
Title: An Open-label, Multi-center Phase I/II Study to Assess the Safety and the Efficacy of SMART101 After Haploidentical Peripheral Blood Stem Transplantation With Post-transplant Cyclophosphamide in Subjects With Hematological Malignancies
Brief Title: Safety and Efficacy of SMART101 in Adult Patients With Hematological Malignancies After Haploidentical HSCT With Post-transplant Cyclophosphamide
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Smart Immune SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SI101-02
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Hematological Malignancies
Keywords: AML, ALL, MSD
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Multiple Sulfatase Deficiency Disease

STUDY DESIGN:
Intervention Model Description: * Phase I/II, open-label, dose-escalation, single arm, multicenter study.
  * This study will comprise two segments:
    * A phase I dose-escalation segment: Three (3) prespecified dose-levels of SMART101 will be evaluated in three consecutive cohorts of patients whatever the type of conditioning regimen the patients will receive before the HSCT to define the SMART101 recommended dose (RecD).
    * A phase II segment: once all patients from the dose-escalation segment have completed their "treatment period " and the SMART101 RecD has been defined, a total number of 34 patients will be enrolled at the RecD in the phase II segment of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with acute leukemia or myelodysplastic syndrome and eligible for an haplo PT-Cy HSCT (Experimental): Segment 1: 3 dose-level SMART101 cells/infusion
  1. 1.5 x 106 CD7+ cells per kg of body weight
  2. 4.5 x 106 CD7+ cells per kg of body weight
  3. 9.0 x 106 CD7+ cells per kg of body weight
  Segment 2:
  2 cohorts of patients will be included in the study based on the type of conditioning regimen:
  * The cohort A will include up to 17 patients receiving a myeloablative conditioning (MAC).
  * The cohort B will include up to 17 patients receiving a reduced intensity conditioning (RIC).
  * Enrollment of patients in each cohort will be done in parallel.
  Interventions: Biological: Allogeneic T cell progenitors, cultured ex-vivo

INTERVENTIONS:
Biological: Allogeneic T cell progenitors, cultured ex-vivo — Injection of T cell progenitors 6 days after haplo HSCT and 2 days after the last administration of cyclophosphamide
  Other Names: SMART101

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of SMART101 (Human T Lymphoid Progenitors (HTLP)) injection to accelerate immune reconstitution after haploidentical hematopoietic stem cell transplantation (HSCT) with post-transplant cyclophosphamide (PT-Cy) in adult patients with hematological malignancies.

ELIGIBILITY:
Main Inclusion Criteria:

* Patients with AML, ALL or MDS eligible for an allogeneic HSCT with a haploidentical donor with post-transplant cyclophosphamide.
* Patients must be ≥ 18 years of age at the time of signing the ICF.
* Patients must have a Karnofsky index ≥ 70%.
* Patients must have a left ventricular ejection fraction of ≥40%.
* Patients must have an intact pulmonary function or Diffusing capacity of the Lungs for Carbon Monoxide (DLCO) ≥ 45% of predicted.
* Patients must have adequate hepatic and renal functions, as assessed by standard laboratory criteria.

Main Exclusion Criteria:

* Patients who have received prior allogeneic stem cell transplantation.
* Patients who have received prior treatment with another cellular therapy within 4 weeks before the planned day of SMART101 infusion.
* Patients who plan to receive, are concurrently receiving or have received any investigational agent within 4 weeks before the planned day of SMART101 infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Unexpected Unacceptable Toxicities (UUT) following the administration of SMART101. | 14 days post SMART101 infusion
  To evaluate the safety of SMART101.
CD4+ T cell count. | 100 days post-HSCT
  to evaluate the efficacy of the study drug

SECONDARY OUTCOMES:
Occurrence of adverse events (AEs) | up to 24 months post-HSCT
T cell immune reconstitution | up to 12 months post-HSCT
  Time course of the T cell immune reconstitution, with a focus on naive CD4+ cells and total CD8+cells
Cumulative incidence of infections | Day 100, and Months 6 and 12 post-HSCT
Non-relapse mortality (NRM) | Day 100, and Months 6, 12 and 24 post-HSCT

OTHER OUTCOMES:
Overall Survival (OS) | Month 24 post-HSCT
Disease-free Survival | Month 24 post-HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Fabio CICERI, MD, Pr., Principal Investigator — I.R.C.C.S. Ospedale San Raffaele
Locations (4):
- France (4):
  - Institut Paoli Calmettes, Marseille
  - Centre hospitalier universitaire de Nantes, Nantes
  - Hôpital Saint-Louis, Paris
  - CHU Toulouse- Institut Universitaire du cancer Toulouse- Oncopole, Toulouse

IPD SHARING:
Plan to Share IPD: No